CLINICAL TRIAL: NCT02166398
Title: Phase 1 Study of Compare the Safety, Pharmacokinetic Profiles of UI15AML055MT and Amosartan® Tablet 5/50 mg
Brief Title: A Randomized, Open-label, Single Dose, Two-way Crossover Clinical Trial to Compare the Safety, Pharmacokinetic Profiles of UI15AML055MT and Amosartan® Tablet 5/50 mg After a Single Oral Administration in Healthy Male Volunteers
Acronym: UI15AML055MT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea United Pharm. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KUP-UNSD-101
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: Amlodipine basylate, Losartan potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amosartan 5/50 tab (Active Comparator): Amosartan 5/50 tab given by oral administration
  Interventions: Drug: Amosartan 5/50
- UI15AML055MT tab (Experimental): UI15AML055MT tab given by oral administration
  Interventions: Drug: UI15AML055MT

INTERVENTIONS:
Drug: UI15AML055MT — tab, PO
  Arms: UI15AML055MT tab
Drug: Amosartan 5/50 — tab, PO
  Arms: Amosartan 5/50 tab

SUMMARY:
A randomized, open-label, single dose, two-way crossover clinical trial to compare the safety, pharmacokinetic profiles of UI15AML055MT and Amosartan® tablet 5/50 mg after a single oral administration in healthy male volunteers

DETAILED DESCRIPTION:
A randomized, open-label, single dose, two-way crossover clinical trial to compare the safety, pharmacokinetic profiles of UI15AML055MT and Amosartan® tablet 5/50 mg after a single oral administration in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Patients over 20 under 45 years of age
* BMI state over 19 under 27

Exclusion Criteria:

* mean sit SBP≥100mmHg or mean sit DBP≥150mmHg at screening
* mean sit SBP≥65mmHg or mean sit DBP≥95mmHg at screening
* Patients showed clinically significant hematological finding, patients with renal diseases (serum creatinine), patients with hepatic disease (ALT or AST)
* History of alcohol or drug abuse
* Positive to pregnancy test, nursing mother, has an intention on pregnancy
* Considered by investigator as not appropriate to participate in the clinical study with othe reason

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
AUClast of Amlodipine | 1d,15d 0h pre-dose, 1, 2, 4, 6, 8, 10, 12, 24, 48, 72, 96, 144h post-dose
AUCinf of Amlodipine | 1d,15d 0h pre-dose, 1, 2, 4, 6, 8, 10, 12, 24, 48, 72, 96, 144h post-dose
Cmax of Amlodipine | 1d,15d 0h pre-dose, 1, 2, 4, 6, 8, 10, 12, 24, 48, 72, 96, 144h post-dose
AUClast of Losartan | 1d,15d 0h pre-dose, 0.25, 0.5, 0.75, 1, 1.25 1.5, 2, 3, 4, 6, 8, 10, 12h post-dose
AUCinf of Losartan | 1d,15d 0h pre-dose, 0.25, 0.5, 0.75, 1, 1.25 1.5, 2, 3, 4, 6, 8, 10, 12h post-dose
Cmax of Losartan | 1d,15d 0h pre-dose, 0.25, 0.5, 0.75, 1, 1.25 1.5, 2, 3, 4, 6, 8, 10, 12h post-dose

SECONDARY OUTCOMES:
Tmax of Amlodipine | 1d,15d 0h pre-dose, 1, 2, 4, 6, 8, 10, 12, 24, 48, 72, 96, 144h post-dose
t1/2 of Amlodipine | 1d,15d 0h pre-dose, 1, 2, 4, 6, 8, 10, 12, 24, 48, 72, 96, 144h post-dose
CL/F of Amlodipine | 1d,15d 0h pre-dose, 1, 2, 4, 6, 8, 10, 12, 24, 48, 72, 96, 144h post-dose
Tmax of Losartan | 1d,15d 0h pre-dose, 0.25, 0.5, 0.75, 1, 1.25 1.5, 2, 3, 4, 6, 8, 10, 12h post-dose
t1/2 of Losartan | 1d,15d 0h pre-dose, 0.25, 0.5, 0.75, 1, 1.25 1.5, 2, 3, 4, 6, 8, 10, 12h post-dose
CL/F of Losartan | 1d,15d 0h pre-dose, 0.25, 0.5, 0.75, 1, 1.25 1.5, 2, 3, 4, 6, 8, 10, 12h post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea